CLINICAL TRIAL: NCT01824069
Title: Phase IIa Clinical Trial to Safety of Treatment in Critical Ischemia Nonrevascularizable Lower Limb by Mesenchymal Stem Cells
Brief Title: Treatment CLI Nonrevascularizable Lower Limb With Cell Therapy
Acronym: HULPVAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HULPVAS-2011-01; 2012-000290-23 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2013-04

CONDITIONS: Nonrevascularizable Critical Ischemia of the Lower Limbs
Keywords: Critical Ischemia; Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous mesenchymal stem cells (Experimental): Intramuscular injection of a suspension of adult mesenchymal stem cells derived from adipose tissue at doses of 1 million per kilo of weight in a dosis
  Interventions: Other: Intramuscular injection of a suspension of adult mesenchymal stem cells derived

INTERVENTIONS:
Other: Intramuscular injection of a suspension of adult mesenchymal stem cells derived — Intramuscular injection of a suspension of adult mesenchymal stem cells derived from adipose tissue at doses of 1 million per kilo of weight. Only one dosis by patients

SUMMARY:
It has been demonstrated the feasibility, safety and effectiveness of mesenchymal stem cells derived from lipoaspirate for treating various pathologies fistula. With this project we will address a study population with critical ischemia of lower limbs without possibility of revascularization, either by technical criteria (no intervention possible to compensate for the lack of irrigation of a limb) criteria or risk / benefit (intolerable surgical risk for the type of intervention required). It will almost always elderly patients with multiple comorbidities and high surgical risk who have a lower limb ischemia in critical degree, with very high probability of major amputation in the short term or immediate.

Hypothesis: mesenchymal stem cells obtained by lipoaspirate expanded "ex vivo", are capable of promoting angiogenesis de novo to improve critical limb ischemia lower nonrevascularizable a safe manner

DETAILED DESCRIPTION:
The primary endpoint of safety and feasibility study will be done when the patient has received treatment at 12 months after implantation. It defines that the process is safe when in the development and monitoring of the trial there has been no adverse events that may be related to the proposed therapy in the trial. All adverse events will be collected during the same time monitoring the clinical evaluation. The main objective will be assessed the cumulative incidence of adverse effects attributed to the study therapy.

Secondary endpoints: As part of the evaluation of the quality of life of patients and clinical evaluation of the treatment will be at 6, 9 and 12 months after implantation a Test SF-12, a magnetic resonance angiography, and tissue oximetry records ankle-brachial index

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent.
2. > 18 years.
3. Chronic arterial ischemia grades IV-V of Rutherford that affects at least one limb.
4. Arterial occlusion direct flow or distal femoropopliteal level.
5. No option for surgical or endovascular revascularization.
6. Life expectancy exceeding two years.
7. High probability of need for major amputation at 6 months (CLI nonrevascularizable).
8. Negative pregnancy test if applicable.

Exclusion Criteria:

1. Background of hematologic neoplasia or unresolved.
2. Hipertensión uncontrolled blood (> 180/110).
3. Severe heart Insuficiencia (New York Heart Association [NYHA] IV) or ejection fraction <30%.
4. Malignant ventricular, Arritmias.
5. Trombosis of deep vein the past three months.
6. active infection.
7. Infarto infarction or stroke the previous three months.
8. Medical or psychiatric illness of any kind which, in the opinion of the investigator, may be a reason for exclusion from the study.
9. Subjects with congenital or acquired immunodeficiencies. Hepatitis B and / or C or tuberculosis diagnosed at the time of inclusion, treponema.
10. Major surgery or severe trauma of the subject in the previous semester.
11. Administration of any investigational drug at present to three months prior to enrollment for this trial.
12. Pulmonary heart disease, in the opinion of the investigator, be unstable or is sufficiently serious to dismiss the patient from the study.
13. Infants or pregnant women.
14. Adult women of childbearing potential not using effective contraception during the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety of inject mesenchymal stem cells in MMII | one year
  It defines that the process is safe when in the development and monitoring of the trial there has been no adverse events that may be related to the proposed therapy in the trial.

SECONDARY OUTCOMES:
Quality of life of patients after treatment | one year
  We analyze the quality of life of patients by SF-12 test

OTHER OUTCOMES:
Clinical evaluation of patients after treatment | One year
  Clinical evaluation of patients after treatment with magnetic resonance angiography, tissue oximetry records and ankle-brachial index.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Riera del Moral, Doctor, Principal Investigator — Instituto de Investigación Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain